CLINICAL TRIAL: NCT03965351
Title: TRPV2 Agonists in Fontan Circulation Patients
Brief Title: TRPV2 Agonists in the Fontan Circulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-0541
Record Dates: First submitted 2018-05-16; First posted 2019-05-29 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-01

CONDITIONS: Fontan
MeSH Terms: interventions — Probenecid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Probenecid (Experimental): the study medication (probenecid) as well as a placebo.
  Interventions: Drug: Probenecid; Other: Placebo
- Placebo (Placebo Comparator): placebo compared to probenecid
  Interventions: Drug: Probenecid; Other: Placebo

INTERVENTIONS:
Drug: Probenecid — This is a cross-over pilot study where participants will receive both the study medication (probenecid), as well as a placebo to see if the study medication improves magnetic resonance parameters of systolic and diastolic dysfunction that occurs in the Fontan population.
Other: Placebo — placebo

SUMMARY:
There are currently very few proven pharmacologic options available for these patients. The recent discovery of transient receptor potential vanilloid (TRPV) channels, particularly TRPV2 channels, in the cardiovascular system is promising as a potential pathway for pharmacologic intervention for Fontan patients. Probenecid, a drug best known as a treatment for gout or as a penicillin adjunct, acts as a TRPV2 agonist and has recently become the subject of study as a model therapy for the treatment of cardiomyopathy due to its positive inotropic and lusitropic effects. The purpose of this pilot study is to determine if probenecid will improve magnetic resonance (MRI) parameters of systolic and/or diastolic dysfunction as well as associated symptoms in patients with a Fontan circulation. The investigators will quantitatively assess functional improvement with pre- and post-treatment cardiopulmonary exercise testing.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 12 years old
2. Single ventricle congenital heart disease status post Fontan procedure.
3. Impaired ventricular function as assessed by preexisting echocardiographic studies and any available MRI studies.

   1. LV inclusion criteria: Ejection fraction by cMRI or echo assessment of <50% or moderate to severe dysfunction.
   2. RV inclusion criteria: Ejection fraction by cMRI of <45% or moderate to severe dysfunction. Or, given the ASE recommendation to avoid use of 2-D imaging quantification for assessment of right ventricular systolic function, a peak global longitudinal strain value as assessed by a single reviewer with a value greater than -17% will also be included. Peak global longitudinal strain analysis will be performed for all eligible single right ventricles noted by subjective echo reports to have abnormal systolic function if no qualifying cardiac MRI assessment of ejection fraction is available.

Exclusion Criteria:

1. Clinically unstable or ongoing illness.
2. Evidence of untreated Fontan pathway obstruction.
3. Presence of uncontrolled arrhythmias.
4. Evidence of moderate or greater atrioventricular valve regurgitation.
5. Pregnancy.
6. History of sulfonamide allergy
7. Known G6PD deficiency
8. Patients on certain drugs that have potentially dangerous interactions with probenecid: doripenem, zalcitabine, deferiperone, citalopram, methotrexate, ciprofloxacin, amoxicillin, cefprozil, cefpodoxime, cefotaxime, meropenem, ertapenem, valganciclovir, ganciclovir, ziovudine ketorolac, cefdinir, cephalexin, dapsone, indomethacin, and piperacillin.Each subject's medication list will be reviewed prior to study participation.
9. Impaired renal function as defined by a GFR < 60mL/min/1.73 m2 within the last year.
10. Patients at a higher risk for arrhythmia including those with a prior history of arrhythmia including atrial and ventricular dysrhythmia or those on established anti-arrhythmic therapy.
11. Admission to the hospital due to a clinically significant arrhythmia within the previous month.
12. Greater than moderate atrioventricular regurgitation as denoted on most recent echo report.
13. Patients with atrio-pulmonary Fontan
14. Currently enrolled in an interventional drug trial or completed an interventional drug trial within the past 30 days.
15. Not appropriate for MRI screening due to having an implanted device.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective randomized, placebo-controlled cross-over pilot study of up to 22 patients who have had a prior Fontan operation for single ventricle physiology who are ≥ 10 years old. Each patient completed a total of four study visits over the course of a 4 month period.
Pre-assignment Details: Each patient came in for a baseline assessment visit. At the end of the baseline visit they received either probenecid or placebo. They took the medication for a month and then returned for the second visit. A washout period occurred for a month and then study patients returned for visit three where they received either probenecid or placebo; whichever was not received during visit one. This medication was taken for a month and then patients returned for the final visit.
Groups:
- Probenecid, and Then Placebo; Placebo, and Then Probenecid: All patients will have a baseline assessment immediately preceding initiation of probenecid or placebo. This will include a physical exam to assess any clinical symptoms, review of cardiac symptoms, blood work, pregnancy test for those girls/women of child bearing potential, PEDS QL questionnaire completion, exercise testing and MRI, as described in detail below. Patients will then receive either probenecid or placebo for 28(±7 days) of treatment according to their randomization group, after which the same testing will be repeated. Following 28(±7 days) of washout, patients will undergo the same testing procedures as during the first period of study but with the alternate treatment. To assist in achieving congruence between clinical testing performed and desired pre-intervention testing, we will coordinate with each patient and his/her cardiologist prior to the clinical visit.
  Patients will receive a one month supply of oral probenecid therapy with the following dosing regimen:
  * For patients (adults and pediatric) ≥ 40 kg: 500 mg by mouth twice daily.
  * For children 10-17 years old and < 40 kg: 250 mg by mouth twice daily
  During the placebo treatment arm, patients will receive 28(±7 days) of placebo therapy. Oral placebo therapy will be twice daily, with an identical dosing regimen as the placebo.
Period: First Intervention (4 Weeks)
Arm/Group | Probenecid, and Then Placebo | Placebo, and Then Probenecid
Started | 3 | 5
Completed | 3 | 4
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Wash Out Period (4 Weeks)
Arm/Group | Probenecid, and Then Placebo | Placebo, and Then Probenecid
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Probenecid, and Then Placebo | Placebo, and Then Probenecid
Started | 3 | 4
Completed | 3 | 3
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Probenecid, Then Placebo: the study medication (probenecid) as well as a placebo.
  Probenecid: This is a cross-over pilot study where participants will receive both the study medication (probenecid), as well as a placebo to see if the study medication improves magnetic resonance parameters of systolic and diastolic dysfunction that occurs in the Fontan population.
  Placebo: placebo
- Placebo, Then Probenecid: placebo compared to probenecid
  Probenecid: This is a cross-over pilot study where participants will receive both the study medication (probenecid), as well as a placebo to see if the study medication improves magnetic resonance parameters of systolic and diastolic dysfunction that occurs in the Fontan population.
  Placebo: placebo
- Total: Total of all reporting groups
Arm/Group | Probenecid, Then Placebo | Placebo, Then Probenecid | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 5 | 8
Left ventricle dominant [Number; unit: participants] | 3 | 5 | 8
Right ventricle dominant [Number; unit: participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in End Diastolic and End Systolic Volume as Measured by Standard and Advanced MRI Parameters
Description: Determine if Fontan patients treated with probenecid for four weeks will experience increased systolic and diastolic function (as measured via standard and advanced MRI parameters) compared with four weeks of placebo. Participants will be assigned to either the placebo arm or study medication arm for the first four weeks. They will then undergo a four week wash out period. Finally, participants will be placed into the study arm that they were not assigned to in the first four weeks when they return for the last four weeks of study participation. There will be four MRI scans over the course of the 12 week study period.
Time Frame: Total time participation in the study will be twelve weeks. Four weeks on the placebo or study medication, four weeks of a washout period and another four weeks with the study medication or placebo.
Measure: Median (Inter-Quartile Range); unit: ml
Groups:
- Probenecid: This is a cross-over pilot study. Results are indicative of subject response when receiving the study medication (probenecid).
- Placebo: This is a cross-over pilot study. Results are indicative of subject response when receiving the placebo medication.
Arm/Group | Probenecid | Placebo
Number analyzed (Participants) | 6 | 6
ml
  End Diastolic Volume | 3.3 [-2.2 to 8.3] | 3.0 [1.1 to 12.1]
  End Systolic Volume | 3.0 [-5.4 to 7.8] | 4.4 [1.8 to 10.9]

2. Secondary Outcome: Changes in Exercise Performance (VO2 Absolute) as Determined by Completing Four Graded Exercise Tests Utilizing a Cycle Ergometer Ramp Protocol; Pre and Post Study Drug and Placebo Administration.
Description: Determine if Fontan patients treated with probenecid for four weeks will experience improved exercise performance compared with four weeks of placebo as measured by a maximal graded exercise test. Participants will complete a graded maximal cycle ergometer test at each of their four study visits.
Time Frame: as for outcome 1
Population: Max VO2 Absolute
Measure: Mean (Inter-Quartile Range); unit: ml/min
Arm/Group | Probenecid | Placebo
Number analyzed (Participants) | 6 | 6
ml/min | 40 [40 to 210] | 70 [10 to 90]

3. Secondary Outcome: Impact of Study Medication on Exercise Capacity (Indexed VO2 [ml/kg/Min] of Single Ventricle Patients.
Description: Determine if there is a quantitative difference in indexed VO2 max when patients have been taking the study medication (probenecid) versus a placebo.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ml/kg/min
Arm/Group | Probenecid | Placebo
Number analyzed (Participants) | 6 | 6
ml/kg/min | 1 [1 to 4] | 1 [1 to 1]

4. Secondary Outcome: Impact of Study Medication on the MRI Ejection Fraction of Single Ventricle Patients.
Description: Determine if there is a quantitative difference in ejection fraction when patients are taking the study medication (probenecid) versus when they are taking a placebo.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent of blood
Arm/Group | Probenecid | Placebo
Number analyzed (Participants) | 6 | 6
percent of blood | -1.2 [-3.1 to 2.7] | -1.1 [-4.0 to 2.6]

5. Secondary Outcome: Impact of Study Medication on MRI Flow Rates of the Ventricles (Cardiac Output) in Single Ventricle Patients
Description: Determine if there is a quantitative difference in cardiac output of single ventricle patients when taking the study medication (probenecid) versus taking a placebo.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: L/min
Arm/Group | Probenecid | Placebo
Number analyzed (Participants) | 3 | 3
L/min | 0.51 [-0.21 to 0.83] | -0.21 [-0.53 to 0.68]

6. Secondary Outcome: Impact of Study Medication on MRI Strain Values in Single Ventricle Patients
Description: Determine if there is a quantitative difference in longitudinal, circumferential, and radial strain MRI values when subjects take the study medication (probenecid) versus a placebo.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Probenecid | Placebo
Number analyzed (Participants) | 6 | 6
percent
  Longitudinal Strain, systole | -2.0 [-3.0 to -2.0] | 1.0 [-1.0 to 2.0]
  Circumferential Strain, systole | 2.0 [-1.0 to 3.0] | -1.0 [-1.0 to 0]
  Radial Strain, systole | 2.5 [-2.0 to 11.0] | 0 [-12.0 to 8.0]
  Longitudinal strain, diastole | 0.14 [0.08 to 0.19] | 0.20 [-1.1 to 0.36]
  Circumferential strain, diastole | -0.23 [-0.31 to 0.02] | 0.10 [-0.44 to 0.68]
  Radial strain, diastole | -0.31 [-1.7 to 1.4] | 0.10 [-2.0 to 0.40]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected on a per patient basis from the beginning of enrollment at consent to subject completion or withdrawal (whichever came first) up to a maximum of 16 weeks
Groups:
- Probenecid: Participants in this arm were randomly assigned to receive probenecid (study medication) during the first phase, then went through a washout phase, and finally received a placebo during the last phase.
- Placebo: Participants in this arm were randomly assigned to receive placebo during the first phase, then went through a washout phase, and finally received the study medication, probenecid, during the last phase.
Arm/Group | Probenecid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 1/8 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probenecid (N=8) | Placebo (N=8)
Contraindicated Medication Taken (Gastrointestinal disorders) | 0 (0) | 1 (1) — Upon medication reconciliation it was determined that a patient had taken a contraindicated medication while enrolled.
Overdose of study medication (Gastrointestinal disorders) | 0 (0) | 1 (1) — One subject, upon medication reconciliation had potentially taken more study medication than indicated due to forgetting if it had already been taken in a given day.
Hospital Admission (Cardiac disorders) | 0 (0) | 1 (1) — Patient admitted for atrial fibrillation. Previous diagnosis of congestive heart failure. Was not taking study medication at time of admission.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probenecid (N=8) | Placebo (N=8)
Sore Throat (General disorders) | 1 (1) | 1 (2)
Loss of appetite (General disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rhinovirus (Immune system disorders) | 1 (2) | 0 (0)
Migraine (General disorders) | 1 (1) | 0 (0)
Weight Gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Elevated NT-proBNP (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT03965351/Prot_SAP_000.pdf